CLINICAL TRIAL: NCT05653791
Title: Intestinal Ultrasonography in Ulcerative Colitis Patients Treated With Filgotinib
Brief Title: Early Intestinal Ultrasound in Predicting Treatment Response to Filgotinib in Ulcerative Colitis
Acronym: STEER
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Galapagos NV (Industry)
Responsible Party: Principal Investigator, Krisztina Gecse, Dr. K.B. Gecse, MD PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: W22_205 # 22.254
Record Dates: First submitted 2022-11-11; First posted 2022-12-16 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Filgotinib treated patients
  Interventions: Diagnostic Test: Intestinal ultrasound

INTERVENTIONS:
Diagnostic Test: Intestinal ultrasound — Ulcerative colitis patients treated with filgotinib will undergo intestinal transabdominal ultrasound at baseline, week 4 and at the time of the follow-up endoscopy (week 10-16)

SUMMARY:
Objective disease assessment in inflammatory bowel diseases at the time of treatment initiation and during follow-up has become gold standard. However, biomarkers, such as C-reactive protein and fecal calprotectin, fail to provide information on disease extent, location or complications. Repeated endoscopic assessments are performed to evaluate mucosal response to treatment, though associated costs, availability, invasiveness and patient preference are considerable limitations. Recently, intestinal ultrasound (IUS) has gained significant momentum as a non-invasive, easily accessible and low-cost alternative for objective assessment. Accordingly, the ECCO-ESGAR guideline recognizes IUS as a potential tool for the diagnosis and for the monitoring of IBD.

Our study aim is to evaluate the change in intestinal ultrasound parameters (as measured by B-mode and SWE at baseline and week 4) to predict endoscopic response and remission as defined by the follow-up endoscopy and measured by the Mayo endoscopic subscore and the UCEIS during treatment with filgotinib

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Endoscopic and/or histological confirmed diagnosis of UC
* UC disease extent proximal to the rectum (ie, left-sided colitis or pancolitis)
* Moderately to severely active UC, defined by an endoscopic Mayo score of ≥ 2
* Indication for receiving filgotinib treatment

Exclusion Criteria:

* Pregnancy
* Inability to give informed consent
* Proctitis only
* Ongoing gastroenteritis
* (Sub)total colectomy
* Obesity (BMI >35 kg/m²)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate to severe UC starting on filgotonib treatment
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the change in intestinal ultrasound parameters to predict endoscopic response as defined by the follow-up endoscopy measured by the Mayo endoscopic subscore during treatment with filgotinib | 10-16 weeks
Evaluate the change in intestinal ultrasound parameters to predict endoscopic response as defined by the follow-up endoscopy and measured by the Ulcerative Colitis Endoscopic Index of Severity (UCEIS) during treatment with filgotinib | 10-16 weeks
Evaluate the change in intestinal ultrasound parameters to predict endoscopic remission as defined by the follow-up endoscopy and measured by the Mayo endoscopic subscore during treatment with filgotinib | 10-16 weeks
Evaluate the change in intestinal ultrasound parameters to predict endoscopic remission as defined by the follow-up endoscopy and measured by the Ulcerative Colitis Endoscopic Index of Severity (UCEIS) during treatment with filgotinib | 10-16 weeks

SECONDARY OUTCOMES:
evaluate the change in IUS parameters (B-mode and shear-wave elastography (SWE; in kPa) at baseline and week 4) to predict clinical response during follow-up endoscopy | 10-16 weeks
  B-mode: bowel wall thickness (BWT), colour doppler signal (CDS), loss of stratification, loss of haustration and presence of lymph nodes
evaluate the change in IUS parameters (B-mode and SWE; measured in kPa) at baseline and week 4) to predict clinical remission during follow-up endoscopy | 10-16 weeks
• to evaluate the change in IUS parameters (as measured by B-mode and SWE at baseline and week 4) to predict biochemical response and remission at the time of the follow-up endoscopy. | 10-16 weeks
• to evaluate the change in IUS parameters (as measured by B-mode and SWE at baseline and week 4) to predict histological remission at the time of the follow-up endoscopy | 10-16 weeks
• to evaluate IUS parameters (as measured in B-mode) in predicting biochemical remission at 1 year (as defined by fecal calprotectin< 150 ug/g) | 52 weeks / 1 year
• to evaluate IUS parameters (as measured in B-mode) in predicting cortico-steroid-free remission at 1 year | 52 weeks / 1 year
• to evaluate IUS parameters (as measured in B-mode) in predicting clinical remission at 1 year (as defined by the Simple Clinical Colitis Activity Index (SCCAI) ≤ 2) | 52 weeks / 1 year
• to evaluate if addition of calprotectin to early IUS (at week 4) could better predict endoscopic response as defined by the follow-up endscopy than IUS or calprotectin alone. | 4 weeks
• to evaluate if addition of calprotectin to early IUS (at week 4) could better predict endoscopic remission as defined by the follow-up endscopy than IUS or calprotectin alone. | 4 weeks
• to evaluate individual wall layer thickness, with special regard to the submucosa, in relation to response to treatment | 10-16 weeks
• to describe SWE (measured in kPa) in patients with moderate to severe UC | 10-16 weeks
• correlate SWE (measured in kPa) with endoscopic findings of disease severity (measured by the Mayo endoscopic subscore) | 10-16 weeks
• correlate SWE (measured in kPa) with endoscopic findings of disease severity (measured by the UCEIS subscore) | 10-16 weeks
• to evaluate correlation between SWE findings and characteristics of the submucosa, including wall layer thickness and hyperechogenicity | 10-16 weeks
• to evaluate the correlation between segmental healing upon endoscopy and IUS | 10-16 weeks

OTHER OUTCOMES:
• Can early (baseline to week 4) changes in IUS parameters (B-mode and SWE) predict long-term clinical (defined by a decrease of ≥ 3 in SCCAI) response at 1 year | between baseline and 52 weeks / 1 year
• Can early (baseline to week 4) changes in IUS parameters (B-mode and SWE) predict long-term clinical (defined by SCCAI ≤ 2) remission at 1 year | between baseline and 52 weeks / 1 year
• Can early (baseline to week 4) changes in IUS parameters predict long-term biochemical response at 1 year (measured by fecal calprotectin <250 µg/g ) | between baseline and 52 weeks / 1 year
• to explore whether early (baseline to week 4) changes in IUS parameters can predict long-term biochemical remission at 1 year (measured by fecal calprotectin <150 µg/g ) | between baseline and 52 weeks / 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, Amsterdam-Zuidoost, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided